CLINICAL TRIAL: NCT02508155
Title: A Randomised, Double-Blind, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MEDI7352 in Subjects With Painful Osteoarthritis of the Knee
Brief Title: A Study of MEDI7352 in Painful Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: D5680C00001
Record Dates: First submitted 2015-07-02; First posted 2015-07-24 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Infusions, Intravenous; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MEDI7352 IV (Experimental): Up to 11 cohorts of subjects are planned to be dosed by IV infusion, with single and multiple ascending doses.
  Interventions: Biological: MEDI7352 for IV infusion
- IV Placebo (Placebo Comparator): Up to 11 cohorts of subjects are planned to be dosed by IV infusion, with single and multiple ascending doses.
  Interventions: Biological: Placebo for IV infusion
- MEDI7352 Subcutaneous Injection (Experimental): 1 cohort of subjects is planned to be dosed by subcutaneous injection, one single ascending dose cohort.
  Interventions: Biological: MEDI7352 for Subcutaneous Injection
- Subcutaneous Placebo (Placebo Comparator): 1 cohort of subjects is planned to be dosed by subcutaneous injection, one single ascending dose cohort.
  Interventions: Biological: Placebo for Subcutaneous Injection

INTERVENTIONS:
Biological: MEDI7352 for IV infusion — MEDI7352 for IV infusion
  Arms: MEDI7352 IV
Biological: Placebo for IV infusion — IV Placebo infusion
  Arms: IV Placebo
Biological: MEDI7352 for Subcutaneous Injection — MEDI7352 for subcutaneous injection
  Arms: MEDI7352 Subcutaneous Injection
Biological: Placebo for Subcutaneous Injection — Subcutaneous Placebo Injection
  Arms: Subcutaneous Placebo

SUMMARY:
The purpose of this study is to assess the safety, drug levels and effects on the body of MEDI7352, in subjects with painful osteoarthritis of the knee.

DETAILED DESCRIPTION:
An interleaved SAD/MAD Study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of MEDI7352 in subjects with painful osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with painful osteoarthritis (OA) of the knee. Female subjects must be postmenopausal or surgically sterile.
* Body weight between 50kg and 145kg
* Willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Current treatment with another biologic therapeutic agent
* Current of historical diagnosis of RA
* Current diagnosis of an immunological condition that is associated with another form of arthritis in addition to OA, including traumatic arthritis or a seronegative spondyloarthropathy
* At risk of destructive arthropathy, including Rapidly Progressive Osteoarthritis (RPOA), osteonecrosis, spontaneous osteonecrosis of the knee, subchondral insufficiency fractures, hip dislocation and pathological fracture
* Presence of clinically significant neuropathy or other clinically significant disorder involving abnormal peripheral sensation.
* Current serious or unstable clinically important illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Adverse events, serious adverse events,
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Clinical laboratory assessments (serum chemistry, hematology, urinalysis)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  12 Lead electrocardiogram (including QTc, QRS, PR intervals and ventricular rate)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Vital signs (systolic and diastolic BP), heart rate
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of MEDI7352 | At screening and at follow up visit.
  MRI

SECONDARY OUTCOMES:
Area under the plasma drug concentration versus time curves for MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Area under the plasma drug concentration versus time curves from zero to infinity and to last observation (AUC 0-inf; AUC 0-t).
Maximum observed plasma drug concentration (Cmax) of MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Maximum observed plasma drug concentration (Cmax).
Time to maximum observed plasma drug concentration (Tmax) of MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Time to maximum observed plasma drug concentration (Tmax).
Terminal plasma elimination half-life (t1/2) of MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Terminal plasma elimination half-life (t1/2).
Apparent clearance (CL/F). | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Apparent clearance (CL/F).
The presence of anti-drug antibodies (ADAs) to MEDI7352 | All visits from screening up to 56 days post single dose/84 days post multiple dose
  The incidence of anti-drug antibodies (a measure of the body's immune response to the drug).
Pain Numerical Rating Scale (NRS) | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Numerical Rating Scale (NRS)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale, stiffness subscale and function subscale. | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale, stiffness subscale and function subscale.
Patients' Global Impression of Change Scale (PGIC) | All visits from screening up to 56 days post single dose/84 days post multiple dose
  Patients' Global Impression of Change Scale (PGIC)

CONTACTS AND LOCATIONS:
Overall Officials: David Bell, MB BCh BAO MRCGP FFPM, Principal Investigator — Biokinetics
Locations (6):
- Research Site, Berlin, Germany
- Sweden (2):
  - Research Site, Göteborg
  - Research Site, Stockholm
- United Kingdom (3):
  - Research Site, Belfast
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home